CLINICAL TRIAL: NCT03344354
Title: InDure: A Clinical Investigation Comparing the In-Use Durability of Double-gloving With Biogel® Surgical Gloves to Three Comparators
Brief Title: Durability of Double-gloving With Biogel® Surgical Gloves When Used by Clinicians/Surgeons
Acronym: InDure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: InDure_G016-002
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Gloves, Surgical

STUDY DESIGN:
Intervention Model Description: This is a non-significant risk, crossover, comparative, prospective, five-armed, open-label clinical investigation in which failure rates of surgical gloves from four manufacturers will be evaluated in double-gloving fashion.
  The investigation is to be conducted over the course of ten (10) periods where the Biogel® brand of NRL and synthetic latex overgloves and undergloves are compared to other brand products from three manufacturers with comparable glove materials and thickness, and used during similar types of procedures. Study clinicians will be divided into five study groups based on specialty: Cardiothoracic and plastic surgery, Neurosurgery, Orthopaedic surgery, Trauma and acute general surgery, and Colorectal surgery. Before the first period each of five study groups will be randomized to one glove brand to start with in period 1. After each period the study group will cross over to the next period and brand of gloves according to a pre-defined order of rotation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Brand 1 (Active Comparator): sterile surgical gloves Two arms of Brand 1 were combined to allow comparison of the total of all comparator gloves.
  Interventions: Device: Biogel
- Brand 2 (Active Comparator): sterile surgical gloves
  Interventions: Device: Ansell
- Brand 3 (Active Comparator): sterile surgical gloves
  Interventions: Device: Cardinal
- Brand 4 (Active Comparator): sterile sergical gloves
  Interventions: Device: Medline

INTERVENTIONS:
Device: Biogel — Sterile surgical gloves used during surgical procedures.
  Arms: Brand 1
Device: Ansell — Sterile surgical gloves used during surgical procedures.
  Arms: Brand 2
Device: Cardinal — Sterile surgical gloves used during surgical procedures.
  Arms: Brand 3
Device: Medline — Sterile surgical gloves used during surgical procedures.
  Arms: Brand 4

SUMMARY:
A prospective open-label study design was chosen because it will provide the most accurate data on the efficacy of four commercially available similar brands of NRL (natural rubber latex) and synthetic latex surgical gloves when they are used for surgeries in a clinical setting. The primary endpoint will be the overall failure rate of the Biogel® sterile surgical undergloves (device) compared to three undergloves brands of surgical gloves. The secondary endpoints are perforation rates of the underglove, the failure rate of the overglove, the frequency of overglove perforation detection by the glove wearer when double-gloving, the ratio of perforations detected of overglove compared to underglove and to determine the frequency of overglove perforation detection by the glove wearer.

The clinical investigation will be statistically powered to test the hypothesis that the failure rate of the Biogel® Sterile Surgical undergloves is different from that of the three comparators.

DETAILED DESCRIPTION:
This is a non-significant risk, cross-over, comparative, prospective, five-armed, open-label clinical investigation in which the perforation rate of surgical gloves from four different manufacturers will be evaluated in double-gloving fashion. Study clinicians who will directly in the sterile field, with a similar surgical procedural work scope will be asked to use gloves from the four manufacturers of surgical gloves while performing surgical procedures. The types of procedures under which the study gloves will be put in use are prosthetic joints arthroplasty and implantation (i.e. orthopedic), trauma surgery, neurosurgery, colorectal and cardiothoracic surgery.

All gloves under evaluation in each phase will be assessed for perforation rate and overall failure on the basis of binomial responses (Y/N) looking at five time points:

* glove failure pre-donning (after removal from pack, prior to donning)
* glove failure during donning (putting the gloves on)
* observed intraoperative glove failure
* glove failure during doffing (glove removal)
* post-procedure: glove perforation and failure determined using a standardized water leak test

No patients have been enrolled in this study therefore no patient data will be assessed.

ELIGIBILITY:
Inclusion Criteria:

All study clinicians, i.e. study glove wearers, must meet all of the following Inclusion Criteria in order to be included in the investigation:

* Must be certified and licensed physician or a clinician in training under supervision in Orthopedic, Neurosurgery, Cardiothoracic, Colorectal or Trauma specialty surgery services or be working in other OR support functions;
* Directly take part in the surgical procedure work within the sterile field;
* Be willing to wear half size larger underglove if recommended by the manufacturer.
* Perform one of the five target procedure groups which is scheduled to last a minimum of 1 hour;
* Be a current employee or active medical staff member with privileges at the institution conducting the clinical investigation;
* Be willing and able to participate in the written user survey and other tasks associated with the clinical investigation and evaluation of the surgical gloves;
* Be willing and able to read, understand and sign the participant information and consent form prior to the initiation of the clinical investigation.

Exclusion Criteria:

All potential study participants who meets any of the following Exclusion Criteria will not be included in the investigation:

* Has had or currently has dermatological or other medical conditions that may prevent proper scrub technique and the use of the sterile study surgical gloves for the duration of the participation in the procedure or the span of time the investigation is to take place;
* Wearing of rings, bracelets, or other jewelry that cannot be removed during glove evaluation;
* Incomplete or absent training on the current clinical investigation plan and study participation responsibilities; and
* Is an employee or staff member of the Sponsor, CRO or any other glove manufacturer; or is an immediate relative of an employee of the Sponsor, CRO or any other glove manufacturer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3507 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Underglove failure rate compared between all competitors | Procedures that are scheduled to last a minimum of one (1) hour long
  To determine and compare the failure rate of the Biogel® natural rubber latex (NRL) and synthetic latex study underglove assortment to all competitors combined as non-Biogel.
Underglove failure rate compared to each of the three comparators | Procedures that are scheduled to last a minimum of one (1) hour long
  To determine and compare the failure rate of the Biogel® natural rubber latex (NRL) and synthetic latex study underglove assortment to each of the three comparators.

SECONDARY OUTCOMES:
Underglove perforation rate compared to each of the three comparators comparators separately and combined as non-Biogel. | Procedures that are scheduled to last a minimum of one (1) hour long
  To determine and compare the perforation rate of the Biogel® NRL and synthetic latex study underglove assortment to that of the three comparators separately and combined as non-Biogel.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Doll, MD, MPH, Principal Investigator — Virginia Commonwealth University Health; Gonzalo M.L. Bearman, Principal Investigator — Virginia Commonwealth University Health
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Doll M, Namoos A, Kang L, Satpathy J, Feldman MJ, Cassano A, Bohl J, Aboutanos MB, Cameron B, Kim J, Asbury C, Haque M, Hess O, Ahlbom H, Bearman G. A randomized trial comparing the intraoperative durability of double-gloving with Biogel(R) surgical gloves to 3 comparators. Antimicrob Steward Healthc Epidemiol. 2024 Oct 10;4(1):e169. doi: 10.1017/ash.2024.431. eCollection 2024. PMID 39430795